CLINICAL TRIAL: NCT03000634
Title: 2015-09: a Phase II Randomized, Open-label Study of Anti-SLAMF7 MAb During Maintenance Therapy Versus Standard Maintenance Therapy in Gene Expression Profiling (GEP)- Defined Low Risk Multiple Myeloma Patients with High Risk Cytogenetic Abnormalities
Brief Title: 2015-09: a Phase II Randomized, Open-label Study of Anti-signaling Lymphocytic Activation Molecule Monoclonal Antibody During Maintenance Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not and will not be initiated due to lack of funding.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 204814
Record Dates: First submitted 2016-12-07; First posted 2016-12-22 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2017-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; Bortezomib; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anti-SLAMF7 mAb+RD alternating every 8 wks with VRD (Experimental): Elotuzumab 10 mg day 1,15 Lenalidomide 25 mg day 1-21 Dexamethasone 20 mg day 1,8,15,22 Bortezomib 1.3 mg day 1,8,15
  Interventions: Drug: Elotuzumab; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- VRD-bortezomib, lenalidomide, dexamethasone (Other): Bortezomib 1.3 mg day 1, 8,15 Lenalidomide 25 mg day 1-21 Dexamethasone 20 mg day 1, 8,15,22
  Interventions: Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Elotuzumab — Administered through a small tube that goes directly into the vein
  Other Names: Elo
  Arms: Anti-SLAMF7 mAb+RD alternating every 8 wks with VRD
Drug: Bortezomib — Administered as a subcutaneous injection under the skin
  Other Names: Velcade
Drug: Lenalidomide — Capsule taken by mouth
  Other Names: Revlimid
Drug: Dexamethasone — Taken by mouth
  Other Names: Decadron

SUMMARY:
This study will compare the effectiveness and safety of maintenance therapy with continuous bortezomib, lenalidomide, and dexamethasone (VRD) compared to maintenance therapy that alternates VRD with Elotuzumab, lenalidomide, and dexamethasone (Elo RD) every eight weeks.

DETAILED DESCRIPTION:
Past studies conducted at the Myeloma Institute have shown that many patients with low-risk disease (as determined by gene array studies - studies that look at specific genes using special equipment) respond very well to treatment. However, about 15% of low-risk patients still relapse during the first three years of treatment, which means that better treatments are still needed.

This study will compare the effectiveness and safety of maintenance therapy with continuous bortezomib, lenalidomide, and dexamethasone (VRD) compared to maintenance therapy that alternates VRD with Elotuzumab, lenalidomide, and dexamethasone (Elo RD) every eight weeks.

Elotuzumab, bortezomib, lenalidomide and dexamethasone are all approved by the FDA for the treatment of patients with multiple myeloma. VRD is the standard maintenance regimen prescribed at the University of Arkansas for Medical Sciences (UAMS) Myeloma Institute for patients with low risk disease. The investigators want to learn if alternating VRD with Elo RD during maintenance therapy will result in better outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age and not older than 75 years of age at the time of enrollment.
* Patients must have completed a Total Therapy-like treatment regimen for newly diagnosed multiple myeloma consisting of induction chemotherapy and stem cell transplant within 4 months of study enrollment. The completed regimen may have also included post-transplant consolidation therapy, but post-transplant consolidation is not required. The regimen must have included, at minimum, a proteasome inhibitor, an immunomodulatory agent, and a corticosteroid.
* Patients must have low-risk disease, defined as an existing myeloma prognostic risk score risk score < 50.4 from a prior bone marrow biopsy sample in which plasma cells were present.
* Patients must have high risk cytogenetic abnormalities, defined as one or more of the following chromosomal aberrations detected by fluorescent in situ hybridization: 17p-, 1q+, t(4;14) and t(14;16).
* Eastern Cooperative Oncology Group ≤ 2, unless solely due to symptoms of multiple myeloma-related bone disease.
* Patients must have absolute neutrophil count(ANC) ≥ 1,000/mm3 and a platelet count of ≥ 100,000/µL, unless lower levels are due to extensive bone marrow plasmacytosis.
* Patients must have a baseline serum creatinine level of < 3 mg/dL and baseline alanine aminotransferase (ALT) < 3x Upper limit of normal (ULN)
* Toxicities related to prior therapies must be resolved to ≤ Grade 2 according to NCI Common Terminology for Adverse Events (CTCAE) Version 4.
* Female patients must be:

  * Postmenopausal for at least 1 year before the screening visit, OR
  * Surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 simultaneous effective methods of contraception, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Male patients, even if surgically sterilized (ie, post-vasectomy) must agree to one of the following:

  * Practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Patients must sign an IRB-approved informed consent indicating their understanding of the proposed treatment and understanding that the protocol has been approved by the Institutional Review Board (IRB).

Exclusion Criteria:

* Female patients who are nursing or pregnant may not participate.
* Women of childbearing potential must have a negative pregnancy documented within one week of beginning study treatment. Refer to the Revlimid Risk Evaluation and Management Strategy (REMS) program for more information.
* History of poorly controlled hypertension, diabetes mellitus, active or uncontrolled hepatitis, or other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol, or that in the opinion of the investigator would constitute a hazard for participating in this study.
* Known Chronic obstructive pulmonary disease with a Forced Expiratory Volume in 1 second (FEV1) less than 50% of predicted normal. Note that FEV1(forced expiratory volume in 1 second) testing is required for patients suspected of having chronic obstructive pulmonary disease.
* Clinically significant cardiac disease, including: myocardial infarction within one year prior to study enrollment or history of unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV); cardiac arrhythmia ≥ Grade 2 or clinical significant electrocardiogram abnormalities.
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment for one year prior to enrollment. Other cancers will be acceptable if the patient's life expectancy exceeds five years.
* Known allergies, hypersensitivity, or intolerance to monoclonal antibodies or human proteins or any of the study medications, their analogues, or excipients in the various formulations of any agent (refer to the latest versions of the package inserts).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients without disease progression within 36 months from start of study treatment. | 36 months
  Progression-Free Survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Faith E Davies, MD, Principal Investigator — University of Arkansas for Medical Science-Myeloma Institute

IPD SHARING:
Plan to Share IPD: No